CLINICAL TRIAL: NCT00492037
Title: A 5-Day, Double-Blind, Placebo-Controlled Multicenter Study of Oral YM087 (CI-1025) to Assess Efficacy and Safety in Patients With Euvolemic or Hypervolemic Hyponatremia
Brief Title: Study of Efficacy & Safety of Oral YM087 in Subjects With Euvolemic or Hypervolemic Hyponatremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Collaborators: Parke-Davis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 087-CL-043; 1025-023
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Hyponatremia
Keywords: hyponatremia; hypervolemic; euvolemic; conivaptan
MeSH Terms: conditions — Hyponatremia | interventions — conivaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: YM087 oral

SUMMARY:
Study of efficacy & safety of oral YM087 in subjects with euvolemic or hypervolemic hyponatremia

ELIGIBILITY:
Inclusion Criteria:

* Serum Sodium 115 to <130mEq/L
* Plasma Osmolarity <290 mOsmol/kg H2O

Exclusion Criteria:

* Significant renal insufficiency
* Serum sodium increase of ≥8 mEq/L over the baseline day ( Hours 0 to 12)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2000-01; Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Change in serum sodium from Baseline Safety of each dosing regimen | Beginning through end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (29):
- Belgium (3):
  - Brussels
  - Liège
  - Tournai
- Finland (2):
  - Jyväskylä
  - Turku
- France (3):
  - Garches
  - Limoges
  - Paris
- Germany (5):
  - Bad Nauheim
  - Berlin
  - Dresdan
  - Göttingen
  - München
- Italy (4):
  - Ferrara
  - Pavia
  - Pisa
  - Verona
- Netherlands (4):
  - Delft
  - Groningen
  - Leiden
  - Nijmegen
- Poland (3):
  - Radomsko
  - Warsaw
  - Wroclaw
- Spain (3):
  - Barcelona
  - Córdoba
  - Madrid
- United Kingdom (2):
  - Cardiff
  - Manchester